CLINICAL TRIAL: NCT03159793
Title: Evaluation of Live Modelling and Filmed Modelling Techniques Versus no Modelling on Child Anxiety During Dental Treatment: A Randomized Clinical Trial
Brief Title: Evaluation of Different Modelling Techniques on Child Anxiety (RCT)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mariam Salah Mohammad Yassin, Principal investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Protocol Paper
Record Dates: First submitted 2017-05-16; First posted 2017-05-19 (Actual); Last update posted 2018-01-25 (Actual); Status verified 2018-01

CONDITIONS: Anxiety
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group A (Active Comparator): Live Modelling
  Interventions: Behavioral: Live Modelling Technique
- Group B (Active Comparator): Filmed Modelling
  Interventions: Behavioral: Filmed Modelling technique
- Group C (No Intervention): No Modelling

INTERVENTIONS:
Behavioral: Live Modelling Technique — Direct observation is the term used to describe both the filmed and live modelling technique. These techniques depend on familiarizing the patient with the dental environment and allowing the patient to ask the questions he/she wants to ask. The patients are shown a film or are permitted to directly observe a cooperative patient undergoing dental treatment. These techniques have no contra indications they simply may be used with any patient.
  Arms: Group A
Behavioral: Filmed Modelling technique — Direct observation is the term used to describe both the filmed and live modelling technique. These techniques depend on familiarizing the patient with the dental environment and allowing the patient to ask the questions he/she wants to ask. The patients are shown a film or are permitted to directly observe a cooperative patient undergoing dental treatment. These techniques have no contra indications they simply may be used with any patient.
  Arms: Group B

SUMMARY:
A huge number of children suffer from anxiety during their dental treatment especially those who did not receive any type of behavior management during their first dental visit. This will result in a more complicated treatment sessions for the children, dentist and the parents. Fear and anxiety control is the key to change the resistant nature of the anxious patients and also allow them to receive the proper treatment they require. From the point of view that there is no difference between the techniques effectiveness, evaluation of two modelling techniques (live modelling and filmed modelling versus no modelling) for children anxious behavior management during the dental treatment will be performed.

DETAILED DESCRIPTION:
i. Diagnosis:

1. History taking [personal, medical and dental].
2. Clinical examination using mirror and probe.
3. Radiographic examination to make sure that the caries is simple.
4. Preoperative photograph is taken.

ii. Interventions to each group

1. Group A: Live modelling technique

   1. In the 1st dental visit the operator will start by measuring the behavior of the child by Frankl behavior rating scale.
   2. A cooperative patient will be the model for the child.
   3. In the 2nd dental visit the pulse oximetry device will be installed on the child's finger and another form of Frankl behavior rating scale is filled.
   4. The treatment is performed as follows:

   i. Place topical anesthesia. ii. Place anesthetic injection. iii. Cavity preparation. iv. Filling material placement. v. Finishing of the filling. e. The child will be asked to complete a facial image scale
2. Group B: video modelling technique (1) In the 1st dental visit the operator will start by measuring the behavior of the child by Frankl behavior rating scale.

   1. A recorded film will be shown to the child.
   2. In the 2nd dental visit the pulse oximetry device will be installed on the child's finger and another form of Frankl behavior rating scale is filled.
   3. The treatment is performed as follows:

   i. Place topical anesthesia. ii. Place anesthetic injection. iii. Cavity preparation. iv. Filling material placement. v. Finishing of the filling. d. The child will be asked to complete a facial image scale.
3. Group C: No modelling

   1. In the 1st dental visit the operator will start by measuring the behavior of the child by Frankl behavior rating scale.
   2. In the 2nd dental visit the pulse oximetry device will be installed on the child's finger and another form to Frankl behavior rating scale.
   3. The treatment is performed as follows:

   i. Place topical anesthesia. ii. Place anesthetic injection. iii. Cavity preparation. iv. Filling material places. v. Finishing of the filling. d. The child will be asked to complete a facial image scale.

ELIGIBILITY:
Inclusion Criteria:

1. English articles
2. In vivo study (RCT)
3. Medically free children
4. Age group 5-6 years old

Exclusion Criteria:

1. Medically compromised children
2. Adult patients

Ages: 5 Years to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 51 (Estimated)
Dates: Start 2017-12-15 (Actual); Primary Completion 2019-03 (Estimated); Study Completion 2019-09 (Estimated)

PRIMARY OUTCOMES:
Dental Anxiety [using Facial Image Scale] | after finishing the procedures in the 2nd dental visit [ after two weeks of allocation]

SECONDARY OUTCOMES:
Oxygen Saturation [using Pulse oximetry] | Readings are taken in the 2nd dental visit [after two weeks from allocation]
Heart Rate [using Pulse oximetry] | Readings are taken in the 2nd dental visit [after two weeks from allocation]
Patient Cooperation [usind Frankl rating scale] | This is perfomred in the allocation visit , in the 1st dental visit [ after a week from allocation], in the 2nd visit [ after two weeks from allocation]

CONTACTS AND LOCATIONS:
Overall Officials: Fatma A El Shehaby, Prof, Study Director — Cairo University; Soad Abd El Moniem, Ass. prof, Study Chair — Cairo University
Locations (1):
- Cairo university, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided